CLINICAL TRIAL: NCT05259969
Title: Energy Availability, Eating Disorder and RED-S Risk, Health Biomarkers, Gut Microbiota Composition and Performance in Competitive Male Athletes Across the Season
Brief Title: Energy Availability in Male Athletes Across the Season
Acronym: EAMAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Nina Mohorko, Principal Investigator, University of Primorska
Other Study IDs: EAMAS
Record Dates: First submitted 2022-01-17; First posted 2022-03-02 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Relative Energy Deficiency in Sport
Keywords: athlete; energy availability; nutrition; eating disorder
MeSH Terms: conditions — Relative Energy Deficiency in Sport; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Serum, Plasma, Stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of proposed cohort observational study is assessing the risk of low energy availability and relative energy deficiency in sport in competitive adult male athletes.

The changes in athlete's energy availability, health biomarkers in blood, gut microbiota composition and performance will be determined in 3 key stages across the season: during preparation, competition and transition period in a subset of athletes.

The study is investigating following specific aims in the cohort of male competitive athletes:

Correlation between energy availability and resting metabolic rate and metabolic functions across the season.

Correlation between energy availability and reproductive functions across the season.

Correlation between energy availability and hematological biomarkers across the season.

Correlation between energy availability and gut microbiota composition across the season.

Correlation between energy availability and performance across the season.

DETAILED DESCRIPTION:
As the initial part of the research the screening for low energy availability, RED-S and eating disorder risk in a larger group of competitive athletes recognized by Olympic Committee of Slovenia will be performed via combination of validated and semi-validated questionnaires: Low Energy Availability in Males Questionnaire, RED-S specific screening tool, Eating Attitude Test (EAT-26) and Eating disorder Inventory - Drive for thinness score.

25 competitive male athletes will be invited for participation in the continuation phase of the research.

Depending on the type of sports, we will define appropriate time intervals for 3 planned laboratory visits. The first visit is planned in the preparation phase, when the workload, given the periodization of the training, is at its peak. The second visit is planned in the competition phase (presumably 6 moths after the 1st visit) and the third one in the transition phase, when the exercise load is the lowest.

The subjects will be informed about the procedure and the aim of the testing prior to its initiation at the introduction meeting. They will be notified about the right to terminate their participation at any moment. Prior to the initiation of the research they will be asked to sign the informed consent form. By doing that they will be informed about the exact procedure regarding how they will be required to keep a 4 day nutrition records with weighted quantities of food and how to keep the log regarding their physical activity. All subjects will be equipped with the acceleration meter.

In the framework of each laboratory visit, the subjects will come fasted, provide a stool sample and fill in the questionnaires, while we will perform anthropometric measurements, resting metabolic rate measurement by using the indirect calorimetry method in draw a venous blood sample. At the end of the visit, participants will undergo a performance test.

ELIGIBILITY:
Inclusion Criteria:

* National Sport Organization identified competitive female or male athlete
* Male athlete actively training for and racing in an Olympic sports event
* Age 18-40 years

Exclusion Criteria:

* Under 15 years old, older than 40 years
* Female
* Para-athlete
* Non active due to illness or injury

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: Olympic Committee of Slovenia recognized (categorized) competitive adult male athletes
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in energy availability among different periods of a season | Through study completion, an average of 1 year.
  Energy intake (kcal/day), energy expenditure (kcal/day) and fat free mass (FFM; kg) will be combined to report energy availability (kcal/kg FFM/day).

SECONDARY OUTCOMES:
Change in resting metabolic rate among different periods of a season | Through study completion, an average of 1 year.
  Resting metabolic rate will be determined with indirect calorimeter and predicted with validated equations and expressed in kJ/day.
Change in body mass among different periods of a season | Through study completion, an average of 1 year.
  Body mass will be measured to the nearest 0.01 kg.
Change in fat free body mass among different periods of a season | Through study completion, an average of 1 year.
  Fat free body mass (FFM [kg]) will be measured with bioelectrical impedance.
Change in percentage of body fat among different periods of a season | Through study completion, an average of 1 year.
  Percentage body fat [%] will be measured with bioelectrical impedance.
Change in iron status markers among different periods of a season | Through study completion, an average of 1 year.
  Serum iron, haemoglobin, ferritin, transferrin and hepcidin concentrations will be measured.
Change in thyroid markers among different periods of a season | Through study completion, an average of 1 year.
  Serum thyroid-stimulating hormone, triiodothyronine and thyroxine concentrations will be measured.
Change in testosteron concentration among different periods of a season | Through study completion, an average of 1 year.
  Serum testosterone concentration will be measured.
Change in cortisol concentration among different periods of a season | Through study completion, an average of 1 year.
  Serum cortisol concentration will be measured.
Change in Low Energy Availability in Males Questionnaire score among different periods of a season | Through study completion, an average of 1 year.
  Low Energy Availability in Males Questionnaire (LEAM-Q) is male-adapted Low Energy Availability in Females Questionnaire by omitting female-speciffic questions. Score range 0-19, higher scores point to higher risk for relative energy deficiency in sport.
Change in Eating Attitude Test-26 score among different periods of a season | Through study completion, an average of 1 year.
  Eating disorder risk will be assessed with Eating Attitude Test (EAT-26). Score range 0-78, higher scores point to higher risk for eating disorder.
Change in Eating disorder Inventory - Drive for thinness score among different periods of a season | Through study completion, an average of 1 year.
  Drive for thinness will be assessed with Eating disorder Inventory- Drive for thinness questionnaire (EDI-DT). Score range 0-21, higher scores point to higher fat phobia.
Change in inflammation markers among different periods of a season | Through study completion, an average of 1 year.
  Serum C-reactive protein and interleukine-6 concentration will be measured.
Change in ghrelin concentration among different periods of a season | Through study completion, an average of 1 year.
  Serum ghrelin concentration will be measured.
Change in growth hormone concentration among different periods of a season | Through study completion, an average of 1 year.
  Serum growth hormone concentration will be measured.
Change in gut microbiota composition among different periods of a season | Through study completion, an average of 1 year.
  Gut microbiota will be analysed from stool samples.
Change in metabolite concentration among different periods of a season | Through study completion, an average of 1 year.
  Serum glucose, lactate and beta-hydroxybutyrate concentrations will be measured.
Change in sport performance among different periods of a season | Through study completion, an average of 1 year.
  Sports specific performance test will be performed.

OTHER OUTCOMES:
Change in lipid profile among different periods of a season | Through study completion, an average of 1 year.
  Serum total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides concentrations will be measured.
Change in leptin concentration among different periods of a season | Through study completion, an average of 1 year.
  Serum leptin concentration will be measured.
Change in insulin-like growth factor 1 concentration among different periods of a season | Through study completion, an average of 1 year.
  Serum Insulin-like growth factor 1 concentration will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Mohorko, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Areta JL, Taylor HL, Koehler K. Low energy availability: history, definition and evidence of its endocrine, metabolic and physiological effects in prospective studies in females and males. Eur J Appl Physiol. 2021 Jan;121(1):1-21. doi: 10.1007/s00421-020-04516-0. Epub 2020 Oct 23. PMID 33095376
- [Background] Burke LM, Lundy B, Fahrenholtz IL, Melin AK. Pitfalls of Conducting and Interpreting Estimates of Energy Availability in Free-Living Athletes. Int J Sport Nutr Exerc Metab. 2018 Jul 1;28(4):350-363. doi: 10.1123/ijsnem.2018-0142. Epub 2018 Jul 20. PMID 30029584
- [Background] Mountjoy M, Sundgot-Borgen JK, Burke LM, Ackerman KE, Blauwet C, Constantini N, Lebrun C, Lundy B, Melin AK, Meyer NL, Sherman RT, Tenforde AS, Klungland Torstveit M, Budgett R. IOC consensus statement on relative energy deficiency in sport (RED-S): 2018 update. Br J Sports Med. 2018 Jun;52(11):687-697. doi: 10.1136/bjsports-2018-099193. No abstract available. PMID 29773536
- [Background] Sim A, Burns SF. Review: questionnaires as measures for low energy availability (LEA) and relative energy deficiency in sport (RED-S) in athletes. J Eat Disord. 2021 Mar 31;9(1):41. doi: 10.1186/s40337-021-00396-7. PMID 33789771
- [Background] Reed JL, De Souza MJ, Williams NI. Changes in energy availability across the season in Division I female soccer players. J Sports Sci. 2013;31(3):314-24. doi: 10.1080/02640414.2012.733019. Epub 2012 Oct 18. PMID 23075047
- [Background] Staal S, Sjodin A, Fahrenholtz I, Bonnesen K, Melin AK. Low RMRratio as a Surrogate Marker for Energy Deficiency, the Choice of Predictive Equation Vital for Correctly Identifying Male and Female Ballet Dancers at Risk. Int J Sport Nutr Exerc Metab. 2018 Jul 1;28(4):412-418. doi: 10.1123/ijsnem.2017-0327. Epub 2018 Jun 22. PMID 29405782
- [Background] Zabriskie HA, Currier BS, Harty PS, Stecker RA, Jagim AR, Kerksick CM. Energy Status and Body Composition Across a Collegiate Women's Lacrosse Season. Nutrients. 2019 Feb 23;11(2):470. doi: 10.3390/nu11020470. PMID 30813399
- [Background] Melin AK, Heikura IA, Tenforde A, Mountjoy M. Energy Availability in Athletics: Health, Performance, and Physique. Int J Sport Nutr Exerc Metab. 2019 Mar 1;29(2):152-164. doi: 10.1123/ijsnem.2018-0201. Epub 2019 Feb 26. PMID 30632422
- [Background] Logue DM, Madigan SM, Melin A, Delahunt E, Heinen M, Donnell SM, Corish CA. Low Energy Availability in Athletes 2020: An Updated Narrative Review of Prevalence, Risk, Within-Day Energy Balance, Knowledge, and Impact on Sports Performance. Nutrients. 2020 Mar 20;12(3):835. doi: 10.3390/nu12030835. PMID 32245088
- [Background] Loucks AB, Kiens B, Wright HH. Energy availability in athletes. J Sports Sci. 2011;29 Suppl 1:S7-15. doi: 10.1080/02640414.2011.588958. Epub 2011 Jul 28. PMID 21793767
- [Background] Mountjoy M, Sundgot-Borgen J, Burke L, Carter S, Constantini N, Lebrun C, Meyer N, Sherman R, Steffen K, Budgett R, Ljungqvist A, Ackerman K. The IOC relative energy deficiency in sport clinical assessment tool (RED-S CAT). Br J Sports Med. 2015 Nov;49(21):1354. No abstract available. PMID 26764434